CLINICAL TRIAL: NCT01649648
Title: Autologous Cord Blood Cells for Hypoxic Ischemic Encephalopathy: Phase I Study of Feasibility and Safety
Brief Title: Autologous Cord Blood Cells for Brain Injury in Term Newborns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRC/EDG/1032/2, EDG09nov061
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2012-04

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic ischemic encephalopathy; Autologous cord blood
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Autologous cord blood cells arm
  Interventions: Biological: Autologous cord blood

INTERVENTIONS:
Biological: Autologous cord blood — Baby's own umbilical cord blood

SUMMARY:
This is a pilot study to test feasibility and safety of collection, preparation and infusion of a baby's own (autologous) umbilical cord blood during the first 3 days of age if the baby is born with signs of brain injury. The cord blood used is fresh (not frozen and then thawed).

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the safety and feasibility of infusions of autologous (the patient's own) umbilical cord blood cells in term gestation newborn infants with hypoxic-ischemic encephalopathy. For this study, infants who have signs of moderate to severe encephalopathy at birth and have cord blood collected at birth can receive their own cord blood cells during the 3 days of age. Babies will be followed for neurodevelopmental outcome at 1, 4 - 6, 9 - 12 months and 18-24 months. MRI brain will be obtained at 1-2 weeks and 4-6 months old.

ELIGIBILITY:
Inclusion Criteria:

1. Autologous umbilical cord blood available
2. >36 weeks gestation
3. Brain injury that satisfies criteria for therapeutic hypothermia
4. Parental informed consent

Exclusion Criteria:

1. Inability to enroll by 3 postnatal days of age.
2. Presence of known chromosomal anomaly.
3. Presence of major congenital anomalies.
4. Severe intrauterine growth restriction
5. Infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist.
6. Parents refuse consent.
7. Attending neonatologist refuses consent.
8. Failure to collect the infant's cord blood and/or laboratory unable to process cord blood

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety | 1-3 days of age
  Adverse event rates occurring in the recipients

SECONDARY OUTCOMES:
Neurodevelopment | 1 month-2 years old
  Peabody tests, Bayley Scales of Infant Development
Brain imaging | 1 week-6 months
  MRI brain at 1-2 weeks old and 4-6 months old

CONTACTS AND LOCATIONS:
Overall Officials: Jiun Lee, MBBS, Principal Investigator — National University Hospital, Singapore; Samuel Rajadurai, MBBS, Principal Investigator — KK Women's and Children's Hospital; Cheo Lian Yeo, MBBS, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No